CLINICAL TRIAL: NCT03156335
Title: Phase I Trial of MR-guided Focused Ultrasound (MRgFUS) Bilateral Capsulotomy for the Treatment of Refractory Obsessive-compulsive Disorder (OCD)
Brief Title: Trial of MR-guided Focused Ultrasound (MRgFUS) Bilateral Capsulotomy for the Treatment of Refractory Obsessive-compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Neurosurgeon, Scientist, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 002-2017
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Focused Ultrasound (Experimental)
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — MR-guided Focused Ultrasound (MRgFUS) offers the possibility of lesioning deep brain targets, while obviating the need for open surgical approaches. There is no radiation, incision, or burr hole, and lesions are generated in real-time under MR image guidance. Intracranial FUS for other applications, essential tremor most notably, has been shown to be safe and effective, recently receiving Health Canada approval for this indication. The technology, methods and procedures used in this study are identical to those in essential tremor.

SUMMARY:
The proposed study is to evaluate the safety and initial efficacy of MRgFUS for patients with treatment-refractory OCD. This study is designed as a prospective, single arm, nonrandomized study. Assessments will be made before and after MRgFUS for adverse events related to treatment, for clinical symptom relief, and quality of life (QoL). The target in the brain chosen for ablation will be the anterior limb of the internal capsule (ALIC) (i.e 'capsulotomy'). Safety will be assessed prospectively in radiologic and clinical terms. Post-procedural imaging will be evaluated for evidence of swelling, hemorrhage, and the evolution of the lesion in the anterior limb of the internal capsule. Patients will be clinically followed up at Day 1, Month 1, Month 3, Month 6 and Month 12 post-procedure. At every follow-up visit, patients will be evaluated for general health, neurological changes, as well as for device/procedure related adverse events. Imaging will also be performed with positron emission tomography (PET) and MRI, as per the Month 3 and Month 12 post-procedure. Feasibility will be evaluated by determining the rate of patient accrual, the tolerability of the procedure for patients, and the technical ability of heating the ALIC to lesional temperatures.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥20 and ≤80 years of age.
2. Patients who are able and willing to give consent and able to attend study visits, as determined by both study Psychiatrist and the surgeon.
3. Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnosis of Obsessive Compulsive Disorder (OCD), at least 5-year illness history with a minimum score of 28 on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS).
4. Medication-refractoriness as determined by an adequate dose and duration of standard psychiatric treatments (including psychotherapy and/or pharmacology) as determined by two psychiatrists associated with the study. Including specifically:

   1. Failed adequate trial of three or more medications accepted as first line in the treatment of OCD
   2. Attempted augmentation, if tolerated, by at least 2 medications known to be first line treatments for OCD
   3. An adequate trial of cognitive behavioural therapy, delivered by a therapist experienced in treating OCD
5. Able to communicate sensations during the ExAblate MRgFUS treatment
6. A consistent dose of all medications in the 30 days prior to study entry.

Exclusion Criteria:

1. Patients with unstable cardiac status [e.g. Unstable angina pectoris on medication, Patients with documented myocardial infarction within six months, Congestive heart failure requiring medication (other than diuretic), Patients on anti-arrhythmic drugs, Severe hypertension (diastolic BP > 100 on medication)]
2. Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
3. Known intolerance or allergies to MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
4. Severely impaired renal function (estimated glomerular filtration rate < 30ml/min/1.73 m2) or receiving dialysis
5. Laboratory biochemical evidence of abnormal bleeding and/or coagulopathy, including risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter or abnormal INR)
6. Cerebrovascular disease (e.g. cerebrovascular accident within 6 months) or history of intracranial hemorrhage
7. Untreated, uncontrolled sleep apnea
8. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
9. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
10. Are participating or have participated in another clinical trial in the last 30 days
11. Patients unable to communicate with the investigator and staff.
12. Presence of significant cognitive impairment
13. Presence of psychosis on clinical evaluation.
14. Patients with brain tumors already known or revealed on pretreatment MRI
15. Currently pregnant (as determined by history and serum HCG) or lactating.
16. Chemical abuse or dependence within the previous six months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 12 months
  Adverse events (AE) will be recorded and categorized according to severity and relationship to procedure

SECONDARY OUTCOMES:
Clinically meaningful reduction in symptoms [Efficacy] | 12 months
  Primary effectiveness will be evaluated using validated scores and subscales related to the symptom being treated (i.e., Yale-Brown Obsessive Compulsive Scale). Efficacy is defined as a clinically meaningful reduction in symptoms at 12 months post-treatment. A patient with OCD is considered to have a treatment response if their YBOCS is reduced by 35% compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD, PhD, Principal Investigator — Sunnybrook Health Sciences Centre, Sunnybrook Research Institute; Zelm Kiss, MD, PhD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothill Medical Centre, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario